CLINICAL TRIAL: NCT04640233
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase II/III Adaptive Clinical Trial to Assess the Safety and Immunogenicity of Gam-COVID-Vac Combined Vector Vaccine for SARS-Сov-2 Infection in Indian Healthy Subjects
Brief Title: Clinical Trial to Assess Safety and Immunogenicity of Gam-COVID-Vac Combined Vector Vaccine for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Сov-2) Infection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other); Russian Direct Investment Fund (Industry); CRO: JSS Medical Research India Pvt. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RDI-GCV-001; CTRI/2020/11/029234 (Other: Clinical Trial Registry of India)
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Prevention
Keywords: Sputnik; Gamaleya
MeSH Terms: interventions — Gam-COVID-Vac vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Group (Experimental): Gam-COVID-Vac combined vector vaccine, 0.5 ml/dose + 0.5 ml/dose prime-boost immunization on day 1 (component I rAd26-S) and on day 21 (component II rAd5-S)
  Interventions: Biological: Gam-COVID-Vac
- Control Group (Placebo Comparator): Placebo, 0.5 ml/dose + 0.5 ml/dose immunization on days 1 and 21
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Gam-COVID-Vac — Vaccine for intramuscular injection
  Arms: Primary Group
Other: Placebo — Placebo comparator
  Arms: Control Group

SUMMARY:
Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Centre Phase II/III Adaptive Clinical Trial to Assess the Safety and Immunogenicity of Gam-COVID-Vac Combined Vector Vaccine for SARS-Сov-2 Infection in Indian Healthy Subjects.

DETAILED DESCRIPTION:
Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Centre Phase II/III Adaptive Clinical Trial to Assess the Safety and Immunogenicity of Gam-COVID-Vac Combined Vector Vaccine for SARS-Сov-2 Infection in Indian Healthy Subjects.

In phase II trial, 100 subjects of immunogenicity group will be enrolled in 3:1 (Test:Placebo) ratio. These 100 subjects will be assessed for safety and immunogenicity outcomes till Day 28 post the first dose of investigational medicinal product (IMP)/placebo administration and will continue with study assessments till Day 180. Safety and immunogenicity data collected till Day 28 will be submitted to the regulatory authority for recommendation to proceed with Phase III recruitment.

In Phase III trial, 1500 subjects will be enrolled and randomized in the ratio of 3:1 (Gam-COVID--Vac : Placebo).

Each subject will participate in this adaptive study phase II/III clinical trial for 180±14 days after the first dose of the IMP/placebo and will have one screening visit and seven on-site visits during the trial period. The IMP/placebo will be administered intramuscularly during vaccination Visits 1 and 3 (Day 1 and Day 21±2). The observation Visits 2, 4, 5, 6, and 7 will be made on Day 19±2, Day 28±2, Day 42±2, Day 90±7, and Day 180±14, respectively. During the observation visits, vital indicators will be assessed in all subjects and changes in the subjects' condition and well being compared to the previous visit will be recorded. The schedule of examination procedures is mentioned in the Schedule of Event tables.

Additionally, the subjects will be able to have remote consultations with the study physician through the weekly telephonic follow-up.

Blood samples will be taken from immunogenicity group of phase II (all 100) and phase III (284 out of 1500) trials during the following visits to assess the immunogenicity parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent of a subject to participate in the trial
2. Males and females aged 18+ years
3. Negative human immunodeficiency virus (HIV 1 & 2) and hepatitis B and C test results
4. Negative immunoglobulin M (IgM) and immunoglobulin G (IgG) SARS-CoV-2 antibodies through enzyme immunoassay test result
5. Negative COVID-2019 Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) test result at the screening visit (72 hours prior to Visit 1 [Day 1])
6. No COVID-2019 in the medical history
7. History of no contact with COVID-2019 persons within at least 14 days before the enrolment (according to subjects)
8. Consent for using effective methods of contraception during the entire trial 1
9. Negative urine pregnancy test at the screening visit (for child-bearing age women)
10. No evident vaccine-induced reactions or complications after receiving immunobiological products in the medical history
11. No acute infectious and/or respiratory diseases within at least 14 days before the enrolment.

Exclusion Criteria:

1. Any vaccination/immunization within 30 days before the enrolment
2. Steroids (except hormonal contraceptives) and immunoglobulins or other blood products therapy not finished 30 days before the enrolment
3. Immunosuppressors therapy finished within 3 months before the enrolment
4. Pregnancy or breast-feeding
5. Acute coronary syndrome or stroke suffered less than one year before the enrolment
6. Tuberculosis, chronic systemic infections
7. Drug allergy (anaphylactic shock, Quincke edema, polymorphic exudative eczema, atopy, serum disease),hypersensitivity or allergic reaction to immunobiological products, known allergic reactions to study product components, acute exacerbation of allergic diseases on the enrolment day
8. Subjects who are on drugs that could have potential drug interactions with adenovirus vaccine
9. Medical history of malignancy
10. Donated blood or plasma (450+ mL) within 2 months before the enrolment
11. Splenectomy in the medical history
12. Neutropenia (absolute neutrophil count less than 1,000 mm3), agranulocytosis, significant blood loss,severe anaemia (haemoglobin less than 80 g/L), immunodeficiency including autoimmune disorders in the medical history within 6 months before the enrolment
13. Active form of a disease caused by the HIV and hepatitis B or C
14. Anorexia, protein deficiency of any origin
15. Tattoos at the injection site (deltoid muscle area), which does not allow assessing the local response to the IMP or placebo administration
16. Alcohol or drug addiction in the medical history.
17. Participation in any other interventional clinical trial within 1 month prior to the Screening
18. Any other medical condition that would limit the participation of the subject as per Investigator discretion
19. Study centre staff or other employees directly involved in the trial and their families
20. Subjects contraindicated for vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | For Phase II study - at Day 28; For Phase III study - till day 180 after first dose
  For Phase II study - - Incidence & severity of adverse events (AEs) after first dose of IMP/Placebo
  For Phase III study -
  - Incidence of related serious adverse events (SAEs) following vaccination during the study
Immunogenicity | For Phase II study - Day 28 after first dose
  For Phase II study -
  - Seroconversion rate of SARS-CoV-2 glycoprotein-specific antibodies in immunogenicity group
Immunogenicity | For Phase III study - Day 42 after first dose
  For Phase III study - Geometric mean titre ratio of SARS-CoV-2 glycoprotein-specific antibodies between IMP and placebo in immunogenicity group

SECONDARY OUTCOMES:
Adverse Events | Baseline to Day 180
  Incidence and severity of adverse events after injecting the first dose of the IMP/placebo
  Incidence of SAE following vaccination
Immunogenicity assessment | Baseline, Day 21, Day 28, Day 42, Day 90, and Day 180
  Seroconversion rate of SARS-CoV-2 glycoprotein-specific antibodies in immunogenicity group
  Seroconversion rate of SARS-CoV-2 virus-neutralizing antibodies in immunogenicity group
Immunogenicity assessment | Baseline, Day 21, Day 28, Day 42, Day 90, and Day 180
  Geometric mean virus-neutralizing antibodies titre in immunogenicity group
Immunogenicity assessment | Baseline, Day 28, Day 42, Day 90 and Day 180
  Interferon gamma concentration in T-cells after restimulation with the SARS-CoV-2 glycoprotein in cell mediated immunogenicity group
Immunogenicity assessment | Baseline, Day 28, Day 42, Day 90 and Day 180
  The number of proliferating cluster of differentiation 4 (CD4) cell and cluster of differentiation 8 (CD8) cells in response to mitogen stimulation in cell mediated immunogenicity group
Percentage of subjects with mild, moderate, severe coronavirus disease 2019 (COVID-19) developed within 6 months after the first dose of the vaccine/placebo | Baseline to Day 180
  Comparing percentage of subjects developing COVID-19 disease between Gam-COVID-Vac combined vector vaccine and placebo based on severity course
Incidence of coronavirus disease 2019 (COVID-19) developed within 6 months after the first dose in trial subjects | Baseline to Day 180
  Comparing incidence of COVID-19 disease between Gam-COVID-Vac combined vector vaccine and placebo

CONTACTS AND LOCATIONS:
Locations (23):
- India (23):
  - S N Medical College, Agra
  - MGM Medical College and Hospital, Aurangabad
  - KLE Prabhakar Kore Hospital, Belagavi
  - Apollo Hospital, Delhi
  - Batra Hospital, Delhi
  - HIMSR with CHRD-SAS, Delhi
  - ESIC Medical College & Hospital, Faridabad
  - AIG hospital, Hyderabad
  - Maharaja Agrasen Superspecialty Hospital, Jaipur
  - GSVM Medical College, Kanpur
  - Peerless Hospital, Kolkata
  - Atharva Hospital, Lucknow
  - St. George's Hospital, Mumbai
  - JSS Hospital, Mysore
  - INCLEN trust and Gurunanak Hospital, Palwal
  - PIMS, Puducherry
  - BJ Sassoon Hospital, Pune
  - KEM Hospital, Pune
  - Noble Hospital Private Limited, Pune
  - BAPS hospital, Sūrat
  - Rhythm Heart Institute, Vadodara
  - Sumandeep Vidyapeeth, Vadodara
  - Christian Medical College, Vellore

IPD SHARING:
Plan to Share IPD: No